CLINICAL TRIAL: NCT00783367
Title: Phase 2 Trial of Lenalidomide (Revlimid)-Dexamethasone + Rituximab in Recurrent Small B-Cell Non-Hodgkin Lymphomas (NHL) Resistant to Rituximab
Brief Title: Combination Therapy Using Lenalidomide (Revlimid)- Low Dose Dexamethasone and Rituximab for Treatment of Rituximab-Resistant, Non-Aggressive B-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02408; UPenn IRB#807684; RV-NHL-PI-0296
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Follicular Lymphoma; Marginal Zone B-Cell Lymphoma; MALT Lymphoma; Lymphoma of Mucosa-Associated Lymphoid Tissue; Lymphoma, Small Lymphocytic; Waldenstrom Macroglobulinemia; Mantle-Cell Lymphoma
Keywords: Revlimid; Celgene brand of lenalidomide; lenalidomide; Rituxan; CD20 antibody, rituximab; rituximab; Follicular Lymphoma; Marginal Zone B-Cell Lymphoma; Lymphoma, Small Lymphocytic; Waldenstrom Macroglobulinemia; Mantle-Cell Lymphoma; Antigens, CD20; refractory; resistantRefractory/progressive lymphoma less than 6 months from first rituximab dose of previous rituximab-containing regimen; Previously treated; Treated with rituximab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenalidomide plus rituximab with dexamethasone (Experimental): Lenalidomide-low dose dexamethasone plus rituximab
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide: 10mg capsules, orally, once daily for each 28 day cycle for the duration of the study
  Other Names: Revlimid (lenalidomide)
Drug: Dexamethasone — Dexamethasone: 8mg tablets, orally, once weekly on days 3, 10, 17, 24 of each 28 day cycle for the duration of the study;
  Other Names: Decadron (dexamethasone)
Drug: Rituximab — Rituximab: 375mg/m2 IV (in the vein), once weekly on days 1, 8, 15, 22 during month 3 of therapy
  Other Names: Rituxan (rituximab)

SUMMARY:
Pre-clinical data and recently published clinical data suggest a synergistic effect between lenalidomide and dexamethasone. We hypothesize that a combination of lenalidomide-dexamethasone can overcome rituximab resistance. To determine the response rate to lenalidomide and dexamethasone plus rituximab therapy in subjects with recurrent small B-cell non-Hodgkin lymphoma who have had lymphoma progression within 6 months of being treated with rituximab alone or with a rituximab-containing regimen, we propose initial treatment with both drugs for two 28-day treatment cycles (Part I). After response assessment following two cycles of lenalidomide-dexamethasone, patients will enter Part II of the study. In Part II, patients will receive lenalidomide-dexamethasone and rituximab to evaluate the potential reversal of rituximab resistance as measured by response to rituximab and progression-free survival following rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated, histologically confirmed follicular lymphoma (grade 1, 2, 3a), marginal zone lymphoma, small lymphocytic lymphoma with less than <5000 lymphocytes/mm3 or lymphoplasmacytic lymphoma with <3g/mL IgM, mantle cell lymphoma by WHO classification
* Flow cytometry or immunohistochemistry must document CD20 antigen expression. Past documentation of CD20 antigen expression is admissible.
* Subjects must have been treated with rituximab in combination with chemotherapy or as monotherapy and must have refractory or progressive disease <6 months from the first rituximab dose of previous rituximab containing regimen
* At least 18 years of age
* ECOG performance status 0-2
* Measurable disease must be present on physical examination or imaging studies. Any tumor mass >2cm is considered measurable.
* Lesions that are considered non-measurable, but assessable include the following: bone lesions, ascites, pleural/pericardial effusion, lymphangitis cutis/pulmonis, bone marrow
* Patients with a history of intravenous drug abuse or any behavior associated with increased risk of HIV infection should be tested for exposure to the HIV virus
* Understand and voluntarily sign an informed consent
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant of ASA may use warfarin or low molecular weight heparin)
* Laboratory test results within these ranges: absolute neutrophil count greater than or equal to 1500/mm3; platelet count greater than or equal to 75,000/mm3; serum creatinine less than or equal to 2.0mg/dL; total bilirubin less than or equal to 1.5mg/dL (unless due to Gilbert's syndrome); AST (SGOT) and ALT (SGPT) less than or equal to 2.5 x ULN or less than or equal to 5 x ULN if hepatic metastases are present
* Disease free of prior malignancies for greater than or equal to 5 years with the exception of currently treated basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from following study procedure
* Pregnant or breast-feeding females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Known positivity for HIV or active infectious Hepatitis, type A, B, or C. Patients who test positive or who are known to be infected are not eligible due to an increased risk of infection with this regimen. HIV testing is not required for study entry, but is required if the patient is perceived to be at risk.
* Known central nervous system involvement by lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2012-11-14 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Schuster, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania; Abramson Cancer Center; Lymphoma Program, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Davis TA, Grillo-Lopez AJ, White CA, McLaughlin P, Czuczman MS, Link BK, Maloney DG, Weaver RL, Rosenberg J, Levy R. Rituximab anti-CD20 monoclonal antibody therapy in non-Hodgkin's lymphoma: safety and efficacy of re-treatment. J Clin Oncol. 2000 Sep;18(17):3135-43. doi: 10.1200/JCO.2000.18.17.3135. PMID 10963642
- [Background] Golay J, Lazzari M, Facchinetti V, Bernasconi S, Borleri G, Barbui T, Rambaldi A, Introna M. CD20 levels determine the in vitro susceptibility to rituximab and complement of B-cell chronic lymphocytic leukemia: further regulation by CD55 and CD59. Blood. 2001 Dec 1;98(12):3383-9. doi: 10.1182/blood.v98.12.3383. PMID 11719378
- [Background] Golay J, Zaffaroni L, Vaccari T, Lazzari M, Borleri GM, Bernasconi S, Tedesco F, Rambaldi A, Introna M. Biologic response of B lymphoma cells to anti-CD20 monoclonal antibody rituximab in vitro: CD55 and CD59 regulate complement-mediated cell lysis. Blood. 2000 Jun 15;95(12):3900-8. PMID 10845926
- [Background] Harjunpaa A, Junnikkala S, Meri S. Rituximab (anti-CD20) therapy of B-cell lymphomas: direct complement killing is superior to cellular effector mechanisms. Scand J Immunol. 2000 Jun;51(6):634-41. doi: 10.1046/j.1365-3083.2000.00745.x. PMID 10849376
- [Background] Smith MR. Rituximab (monoclonal anti-CD20 antibody): mechanisms of action and resistance. Oncogene. 2003 Oct 20;22(47):7359-68. doi: 10.1038/sj.onc.1206939. PMID 14576843
- [Background] Hofmeister JK, Cooney D, Coggeshall KM. Clustered CD20 induced apoptosis: src-family kinase, the proximal regulator of tyrosine phosphorylation, calcium influx, and caspase 3-dependent apoptosis. Blood Cells Mol Dis. 2000 Apr;26(2):133-43. doi: 10.1006/bcmd.2000.0287. PMID 10753604
- [Background] Clynes RA, Towers TL, Presta LG, Ravetch JV. Inhibitory Fc receptors modulate in vivo cytotoxicity against tumor targets. Nat Med. 2000 Apr;6(4):443-6. doi: 10.1038/74704. PMID 10742152
- [Background] Cartron G, Dacheux L, Salles G, Solal-Celigny P, Bardos P, Colombat P, Watier H. Therapeutic activity of humanized anti-CD20 monoclonal antibody and polymorphism in IgG Fc receptor FcgammaRIIIa gene. Blood. 2002 Feb 1;99(3):754-8. doi: 10.1182/blood.v99.3.754. PMID 11806974
- [Background] Weng WK, Levy R. Two immunoglobulin G fragment C receptor polymorphisms independently predict response to rituximab in patients with follicular lymphoma. J Clin Oncol. 2003 Nov 1;21(21):3940-7. doi: 10.1200/JCO.2003.05.013. Epub 2003 Sep 15. PMID 12975461
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] van der Kolk LE, Grillo-Lopez AJ, Baars JW, Hack CE, van Oers MH. Complement activation plays a key role in the side-effects of rituximab treatment. Br J Haematol. 2001 Dec;115(4):807-11. doi: 10.1046/j.1365-2141.2001.03166.x. PMID 11843813
- [Background] Alas S, Emmanouilides C, Bonavida B. Inhibition of interleukin 10 by rituximab results in down-regulation of bcl-2 and sensitization of B-cell non-Hodgkin's lymphoma to apoptosis. Clin Cancer Res. 2001 Mar;7(3):709-23. PMID 11297268
- [Background] Bohen SP, Troyanskaya OG, Alter O, Warnke R, Botstein D, Brown PO, Levy R. Variation in gene expression patterns in follicular lymphoma and the response to rituximab. Proc Natl Acad Sci U S A. 2003 Feb 18;100(4):1926-30. doi: 10.1073/pnas.0437875100. Epub 2003 Feb 5. PMID 12571354
- [Background] Dave SS, Wright G, Tan B, Rosenwald A, Gascoyne RD, Chan WC, Fisher RI, Braziel RM, Rimsza LM, Grogan TM, Miller TP, LeBlanc M, Greiner TC, Weisenburger DD, Lynch JC, Vose J, Armitage JO, Smeland EB, Kvaloy S, Holte H, Delabie J, Connors JM, Lansdorp PM, Ouyang Q, Lister TA, Davies AJ, Norton AJ, Muller-Hermelink HK, Ott G, Campo E, Montserrat E, Wilson WH, Jaffe ES, Simon R, Yang L, Powell J, Zhao H, Goldschmidt N, Chiorazzi M, Staudt LM. Prediction of survival in follicular lymphoma based on molecular features of tumor-infiltrating immune cells. N Engl J Med. 2004 Nov 18;351(21):2159-69. doi: 10.1056/NEJMoa041869. PMID 15548776
- [Background] Witzig TE, Flinn IW, Gordon LI, Emmanouilides C, Czuczman MS, Saleh MN, Cripe L, Wiseman G, Olejnik T, Multani PS, White CA. Treatment with ibritumomab tiuxetan radioimmunotherapy in patients with rituximab-refractory follicular non-Hodgkin's lymphoma. J Clin Oncol. 2002 Aug 1;20(15):3262-9. doi: 10.1200/JCO.2002.11.017. PMID 12149300
- [Background] Ansell SM, Ristow KM, Habermann TM, Wiseman GA, Witzig TE. Subsequent chemotherapy regimens are well tolerated after radioimmunotherapy with yttrium-90 ibritumomab tiuxetan for non-Hodgkin's lymphoma. J Clin Oncol. 2002 Sep 15;20(18):3885-90. doi: 10.1200/JCO.2002.10.143. PMID 12228209
- [Background] Davis TA, Maloney DG, Grillo-Lopez AJ, White CA, Williams ME, Weiner GJ, Dowden S, Levy R. Combination immunotherapy of relapsed or refractory low-grade or follicular non-Hodgkin's lymphoma with rituximab and interferon-alpha-2a. Clin Cancer Res. 2000 Jul;6(7):2644-52. PMID 10914705
- [Background] Friedberg JW, Kim H, McCauley M, Hessel EM, Sims P, Fisher DC, Nadler LM, Coffman RL, Freedman AS. Combination immunotherapy with a CpG oligonucleotide (1018 ISS) and rituximab in patients with non-Hodgkin lymphoma: increased interferon-alpha/beta-inducible gene expression, without significant toxicity. Blood. 2005 Jan 15;105(2):489-95. doi: 10.1182/blood-2004-06-2156. Epub 2004 Sep 9. PMID 15358617
- [Background] Gluck WL, Hurst D, Yuen A, Levine AM, Dayton MA, Gockerman JP, Lucas J, Denis-Mize K, Tong B, Navis D, Difrancesco A, Milan S, Wilson SE, Wolin M. Phase I studies of interleukin (IL)-2 and rituximab in B-cell non-hodgkin's lymphoma: IL-2 mediated natural killer cell expansion correlations with clinical response. Clin Cancer Res. 2004 Apr 1;10(7):2253-64. doi: 10.1158/1078-0432.ccr-1087-3. PMID 15073100
- [Background] Hernandez-Ilizaliturri FJ, Reddy N, Holkova B, Ottman E, Czuczman MS. Immunomodulatory drug CC-5013 or CC-4047 and rituximab enhance antitumor activity in a severe combined immunodeficient mouse lymphoma model. Clin Cancer Res. 2005 Aug 15;11(16):5984-92. doi: 10.1158/1078-0432.CCR-05-0577. PMID 16115943
- [Background] Wu L, Adams M, Carter T, Chen R, Muller G, Stirling D, Schafer P, Bartlett JB. lenalidomide enhances natural killer cell and monocyte-mediated antibody-dependent cellular cytotoxicity of rituximab-treated CD20+ tumor cells. Clin Cancer Res. 2008 Jul 15;14(14):4650-7. doi: 10.1158/1078-0432.CCR-07-4405. PMID 18628480
- [Background] Reddy N, Hernandez-Ilizaliturri FJ, Deeb G, Roth M, Vaughn M, Knight J, Wallace P, Czuczman MS. Immunomodulatory drugs stimulate natural killer-cell function, alter cytokine production by dendritic cells, and inhibit angiogenesis enhancing the anti-tumour activity of rituximab in vivo. Br J Haematol. 2008 Jan;140(1):36-45. doi: 10.1111/j.1365-2141.2007.06841.x. Epub 2007 Nov 9. PMID 17995965
- [Background] Chanan-Khan A, Miller KC, Musial L, Lawrence D, Padmanabhan S, Takeshita K, Porter CW, Goodrich DW, Bernstein ZP, Wallace P, Spaner D, Mohr A, Byrne C, Hernandez-Ilizaliturri F, Chrystal C, Starostik P, Czuczman MS. Clinical efficacy of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase II study. J Clin Oncol. 2006 Dec 1;24(34):5343-9. doi: 10.1200/JCO.2005.05.0401. Epub 2006 Nov 6. PMID 17088571

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Revlimid + rituximab with dexamethasone
- Cohort 2: Revlimid + rituximab (without dexamethasone)
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 00 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 15 | 19 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to Lenalidomide-dexamethasone + Rituximab Therapy in Relapsed Small B-cell Lymphoma With Rituximab Resistance
Description: Response rate is defined as a complete response or partial response using anatomic criteria of the International Workshop Response Critieria (Cheson, 1999).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 24 | 19
Participants | 14 | 13

2. Secondary Outcome: Time Until Progression After Lenalidomide-dexamethasone + Rituximab Therapy in Relapsed Small B-cell Lymphomas With Rituximab Resistance
Description: Progression free survival time in months
Time Frame: 9 years from enrollment of first subject
Population: Subjects who received both Revlimid and rituximab were evaluable for response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 26 | 19
months | 22.2 [11.4 to 60.8] | 22.4 [7.7 to 30.1]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for each subject from time of start of study therapy through 30 days following last dose of study therapy. Results reported here reflect 15 months following the start of the final subject on study therapy
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 3/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 12/27 | 9/23
Other Adverse Events (participants affected / at risk) | 27/27 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=27) | Cohort 2 (N=23)
Neutrophil count decreased (Investigations) | 2 (3) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
lung infection (Infections and infestations) | 1 (1) | 0 (0) — pneumonia
fever (General disorders) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions, other: tumor flare (General disorders) | 0 (0) | 1 (1) — Tumor Flare
Neoplasms benign, malignant, and unspecified, Other: unrelated second malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) — unrelated second malignancies
Pelvic Infection (Infections and infestations) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infections and infestations - Other: infection of aerodigestive tract (Infections and infestations) | 1 (1) | 0 (0) — Infection of aerodigestive tract
allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — with cardiac ischemia
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=27) | Cohort 2 (N=23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 6 | 9
Constipation (Gastrointestinal disorders) | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Myalgias (Musculoskeletal and connective tissue disorders) | 9 | 7
Diarrhea (Gastrointestinal disorders) | 9 | 10
Fatigue (General disorders) | 20 | 12
dyspepsia (Gastrointestinal disorders) | 4 | 2
hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 6 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Platelet count decreased (Investigations) | 3 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 8
stomach pain (Gastrointestinal disorders) | 0 | 2
General disorders and administration site conditions, other: tumor flare (General disorders) | 4 | 5
Dysgeusia (Nervous system disorders) | 2 | 0
Skin and subcutaneous tissue disorders, other: erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 10 | 0
Lung infection (Infections and infestations) | 3 | 0 — pneumonia
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Weight loss (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT00783367/Prot_SAP_000.pdf